CLINICAL TRIAL: NCT05587725
Title: A Cross-sectional Study to Evaluate the Prevalence of HPV in Gay and Bisexual Men Aged 16-20 Years in Australia
Brief Title: Human Papillomavirus in Young People Epidemiological Research 3
Acronym: HYPER3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Monash University (Other)
Collaborators: The Alfred (Other); University of Melbourne (Other)
Responsible Party: Principal Investigator, Eric Chow, Associate Professor, Monash University
Other Study IDs: 14/22
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Human Papillomavirus Infection; HPV; HPV Infection; Anal Cancer; Cancer; Men; HPV 16 Infection
Keywords: Vaccination; Vaccine; Public health; Prevention; Men who have sex with men; Gay and bisexual men; Immunisation
MeSH Terms: conditions — Papillomavirus Infections; Anus Neoplasms; Neoplasms; Multiple Endocrine Neoplasia Type 1; Homosexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. Self-collected oral rinse sample for HPV testing
  2. Self-collected penile swab for HPV testing
  3. Clinician-collected anal swab for HPV testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anal cancer is overrepresented among gay, bisexual and other men who have sex with men (MSM), particularly those living with HIV. Australia was the first country to introduce a publicly funded national HPV vaccination program in 2007. This program was expanded to include schoolboys aged 12-13 years in 2013; with a 2-year catch-up for boys aged up to 15 years. In 2018, the 9-valent vaccine (covering genotypes 6/11/16/18/31/33/45/52/58) replaced the 4-valent vaccine in the national program.

The goal of the HYPER3 study is to determine the prevalence of anal, genital and oral HPV among 200 young gay and bisexual men aged 16-20 years who were eligible for the school-based 9-valent vaccination.

Participants will be required to complete a questionnaire and provide samples for HPV testing. No follow-up visits will be required.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 16 to 20 (i.e. men aged 16-18 years in 2023; men aged 16-19 years in 2024; and men aged 16-20 years in 2025 will be recruited. This is to ensure these men would have been eligible for the 9-valent school-based HPV program)
* Same-sex attracted
* Residing in Australia since 2018

Exclusion Criteria:

* Unable to complete all study requirements in English

Ages: 16 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Study participants will be recruited from sexual health clinics, community, gay community events, universities, social networking services, and peer-referral.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of quadrivalent vaccine HPV types | Baseline
  The oral, penile and anal prevalence of quadrivalent vaccine types (6, 11, 16 and 18)
Prevalence of nonavalent vaccine HPV types | Baseline
  The oral, penile and anal prevalence of nonavalent vaccine types (6, 11, 16, 18, 31,33, 45, 52 and 58)
Prevalence of type-specific HPV types | Baseline
  The oral, penile and anal prevalence of type-specific HPV types

CONTACTS AND LOCATIONS:
Locations (1):
- Melbourne Sexual Health Centre, Melbourne, Victoria, Australia